CLINICAL TRIAL: NCT01546038
Title: A PHASE 1B/2 STUDY TO EVALUATE THE SAFETY AND EFFICACY OF PF-04449913, AN ORAL HEDGEHOG INHIBITOR, IN COMBINATION WITH INTENSIVE CHEMOTHERAPY, LOW DOSE ARA-C OR DECITABINE IN PATIENTS WITH ACUTE MYELOID LEUKEMIA OR HIGH-RISK MYELODYSPLASTIC SYNDROME
Brief Title: A Study To Evaluate PF-04449913 With Chemotherapy In Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: B1371003; 2012-000684-24 (EudraCT Number)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Hedgehog Inhibitor; Acute Myeloid Leukemia; Myelodysplastic syndrome; Intensive chemotherapy; LDAC; glasdegib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — glasdegib; Cytarabine; Decitabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm A (Phase 1B) (Experimental): PF-04449913 in combination with low dose ARA-C (LDAC)
  Interventions: Drug: PF-04449913; Drug: Low dose ARA-C (LDAC)
- Arm B (Phase 1B) (Experimental): PF-04449913 in combination with Decitabine
  Interventions: Drug: PF-04449913; Drug: Decitabine
- Arm C (Phase 1B) (Experimental): PF-04449913 in combination with intensive chemotherapy: PF-04449913 administered continuously for 28 days. Daunorubicin given using 60 mg/m2 for 3-days together with cytarabine 100 mg/m2 on days 1 through 7 followed by cytarabine 1g/m2 on days 1, 3, and 5 during 2-4 cycles of consolidation therapy.
  Interventions: Drug: PF-04449913; Drug: Daunorubicin; Drug: Cytarabine
- P2 Fit (Phase 2 Single Arm) (Experimental): PF-04449913 in combination with intensive chemotherapy: PF-04449913 administered continuously for 28 days. Daunorubicin given using 60 mg/m2 for 3-days together with cytarabine 100 mg/m2 on days 1 through 7 followed by cytarabine 1g/m2 on days 1, 3, and 5 during 2-4 cycles of consolidation therapy.
  Interventions: Drug: PF-04449913; Drug: Daunorubicin; Drug: Cytarabine
- P2 Unfit (Phase 2 Randomized) (Other): Patients will be randomized 2:1 (low dose ARA-C in combination with PF-04449913: low dose ARA-C alone).
  Interventions: Drug: PF-04449913; Drug: Low dose ARA-C (LDAC)

INTERVENTIONS:
Drug: PF-04449913 — PF-04449913 administered orally and continuously for 28-days.
  Arms: Arm A (Phase 1B)
Drug: Low dose ARA-C (LDAC) — Low dose ARA-C (LDAC) administered at 20 mg SQ, BID on Days 1 through 10.
  Arms: Arm A (Phase 1B)
Drug: PF-04449913 — PF-04449913 administered orally and continuously for 28 days.
  Arms: Arm B (Phase 1B)
Drug: Decitabine — Decitabine given at 20 mg/m2 over 1 hour infusion for 5-days
  Arms: Arm B (Phase 1B)
Drug: PF-04449913 — PF-04449913 administered orally and continuously for 28 days
  Arms: Arm C (Phase 1B)
Drug: Daunorubicin — Daunorubicin given using 60 mg/m2 for 3-days
  Arms: Arm C (Phase 1B)
Drug: Cytarabine — Cytarabine 100 mg/m2 on days 1 through 7
  Arms: Arm C (Phase 1B)
Drug: PF-04449913 — PF-04449913 administered orally and continuously for 28 days
  Arms: P2 Fit (Phase 2 Single Arm)
Drug: Daunorubicin — Daunorubicin given using 60 mg/m2 for 3-days
  Arms: P2 Fit (Phase 2 Single Arm)
Drug: Cytarabine — Cytarabine 100 mg/m2 on days 1 through 7
  Arms: P2 Fit (Phase 2 Single Arm)
Drug: PF-04449913 — PF-04449913 administered orally and continuously for 28 days (if randomized to receive PF-04449913)
  Arms: P2 Unfit (Phase 2 Randomized)
Drug: Low dose ARA-C (LDAC) — Low dose ARA-C (LDAC) administered at 20 mg SQ, BID on Days 1 through 10.
  Arms: P2 Unfit (Phase 2 Randomized)

SUMMARY:
This is a study to evaluate PF-04449913 (an inhibitor of the Hedgehog pathway) in Acute Myeloid Leukemia and high-risk Myelodysplastic Syndrome in combination with standard agents used to treat these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML or RAEB 2 High Risk MDS who are newly diagnosed according to the WHO 2008 Classification and previously untreated.
* Patients with AML (arising from an antecedent hematologic disease [AHD]) or MDS who may have had one prior regimen with commercially available agents for the treatment of their prior hematologic disease. The patients may not have had a prior therapy for their AML.
* AML patients include de novo AML, AML evolving from MDS or other AHD and AML after previous cytotoxic therapy or radiation (secondary AML)
* For a diagnosis of AML, a bone marrow blast count of 20% or more is required.
* For a diagnosis of high-risk Myelodysplastic Syndrome RAEB 2 the patient must have 10-19% bone marrow blasts
* Adequate Organ Function
* ECOG Performance Status 0, 1, or 2

Exclusion Criteria:

* AML M3 Acute Promyelocytic Leukemia (APL) or patients with a t(9:22) cytogenetic translocation.
* Patients with known active uncontrolled central nervous system (CNS) leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2012-06-27 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (79):
- United States (50):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC San Diego Moores Cancer Center - Investigational Drug Services, La Jolla, California
  - UC San Diego Medical Center - La Jolla, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC & USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center / Investigational Drug Services, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center Drug Information Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Drug lnformation/lnvestigational Drugs, Los Angeles, California
  - UCLA Hematology/Oncology Clinic, Los Angeles, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - H.Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service, Emory University Clinic, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Medicine Developmental Therapeutics Institute, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - The University of Chicago's Medical Center, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Clinical Trials Office, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes Jewish Hospital North Campus, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine - Division of Bone Marrow Transplant & Leukemia, St Louis, Missouri
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic Cancer Institute, Cleveland, Ohio
  - Centennial Medical Center, Nashville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Canada (2):
  - Juravinski Cancer Centre @ Hamilton Health Sciences, Hamilton, Ontario
  - Centre de Sante et de Services Sociaux (CSSS) Champlain - Charles-Le Moyne, Greenfield Park, Quebec
- Germany (11):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Johann Wolfgang Goethe University, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Charite -Universitatsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charite - Universitatsmedizin Berlin, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universitaetsklinikum Magdeburg A.oe.R., Magdeburg
  - Johannes Gutenberg-Universitaet Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinikum Ulm, Ulm
- Italy (5):
  - Policlinico S. Orsola-Malpighi, Bologna, Province of Bologna
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Policlinico Universitario "Umberto I" Universita degli Studi "La Sapienza" Sezione di Ematologia, Rome
  - A.O. Citta della Salute e della Scienza di Torino - S.C. Ematologia, Torino
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne Gdanskiego Uniwersytetu Medycznego, Gdansk, Pomeranian Voivodeship
  - Oddzial Hematologii Z pododzialem chemioterapii-Klinika Hematologii Wojewodzkie Wielospecjalistyczne, Lodz
  - Dolnoslaskie Centrum Transplantacji Komorkowych z Krajowym Bankiem Dawcow Szpiku, Wroclaw
- Spain (8):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Heuser M, Smith BD, Fiedler W, Sekeres MA, Montesinos P, Leber B, Merchant A, Papayannidis C, Perez-Simon JA, Hoang CJ, O'Brien T, Ma WW, Zeremski M, O'Connell A, Chan G, Cortes JE. Clinical benefit of glasdegib plus low-dose cytarabine in patients with de novo and secondary acute myeloid leukemia: long-term analysis of a phase II randomized trial. Ann Hematol. 2021 May;100(5):1181-1194. doi: 10.1007/s00277-021-04465-4. Epub 2021 Mar 19. PMID 33740113
- [Derived] Lin S, Shaik N, Chan G, Cortes JE, Ruiz-Garcia A. An evaluation of overall survival in patients with newly diagnosed acute myeloid leukemia and the relationship with glasdegib treatment and exposure. Cancer Chemother Pharmacol. 2020 Oct;86(4):451-459. doi: 10.1007/s00280-020-04132-x. Epub 2020 Sep 3. PMID 32885274
- [Derived] Cortes JE, Heidel FH, Fiedler W, Smith BD, Robak T, Montesinos P, Candoni A, Leber B, Sekeres MA, Pollyea DA, Ferdinand R, Ma WW, O'Brien T, O'Connell A, Chan G, Heuser M. Survival outcomes and clinical benefit in patients with acute myeloid leukemia treated with glasdegib and low-dose cytarabine according to response to therapy. J Hematol Oncol. 2020 Jul 14;13(1):92. doi: 10.1186/s13045-020-00929-8. PMID 32664995
- [Derived] Cortes JE, Heidel FH, Hellmann A, Fiedler W, Smith BD, Robak T, Montesinos P, Pollyea DA, DesJardins P, Ottmann O, Ma WW, Shaik MN, Laird AD, Zeremski M, O'Connell A, Chan G, Heuser M. Randomized comparison of low dose cytarabine with or without glasdegib in patients with newly diagnosed acute myeloid leukemia or high-risk myelodysplastic syndrome. Leukemia. 2019 Feb;33(2):379-389. doi: 10.1038/s41375-018-0312-9. Epub 2018 Dec 16. PMID 30555165
- [Derived] Cortes JE, Douglas Smith B, Wang ES, Merchant A, Oehler VG, Arellano M, DeAngelo DJ, Pollyea DA, Sekeres MA, Robak T, Ma WW, Zeremski M, Naveed Shaik M, Douglas Laird A, O'Connell A, Chan G, Schroeder MA. Glasdegib in combination with cytarabine and daunorubicin in patients with AML or high-risk MDS: Phase 2 study results. Am J Hematol. 2018 Nov;93(11):1301-1310. doi: 10.1002/ajh.25238. Epub 2018 Sep 9. PMID 30074259
- [Derived] Savona MR, Pollyea DA, Stock W, Oehler VG, Schroeder MA, Lancet J, McCloskey J, Kantarjian HM, Ma WW, Shaik MN, Laird AD, Zeremski M, O'Connell A, Chan G, Cortes JE. Phase Ib Study of Glasdegib, a Hedgehog Pathway Inhibitor, in Combination with Standard Chemotherapy in Patients with AML or High-Risk MDS. Clin Cancer Res. 2018 May 15;24(10):2294-2303. doi: 10.1158/1078-0432.CCR-17-2824. Epub 2018 Feb 20. PMID 29463550
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371003&StudyName=A%20Study%20To%20Evaluate%20PF-04449913%20With%20Chemotherapy%20In%20Patients%20With%20Acute%20Myeloid%20Leukemia%20or%20Myelodysplastic%20Syndrome%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1B:Unfit(unfit for intensive chemotherapy)participants with prior decitabine or azacitidine for high risk MDS or AHD(antecedent hematologic disease)were eligible for the LDAC arm only;with prior cytarabine were eligible for decitabine arm only.Phase 2:Participant's treatment arm assignment was based on the fit or unfit status at screening.
Groups:
- Phase 1B: Glasdegib 100 mg + LDAC: Participants received oral doses of glasdegib (PF-04449913) tablets 100 milligram (mg) starting on Day 3 of Cycle 1 for pharmacokinetic (PK) assessment purposes and thereafter once daily (QD) and continuously for 28-day cycles (starting on Day 1 for all other cycles). Low dose Ara-C (LDAC) was given at a dose of 20 mg subcutaneously twice daily (BID) on Days 1-10 of the 28-day cycles.
- Phase 1B: Glasdegib 200 mg + LDAC: Participants received oral doses of glasdegib tablets 200 mg starting on Day 3 of Cycle 1 for PK assessment purposes and thereafter QD and continuously for 28-day cycles (starting on Day 1 for all other cycles). LDAC was given at a dose of 20 mg subcutaneously BID on Days 1-10 of the 28-day cycles. In March 2013, all active participants receiving glasdegib 200 mg were required to reduce dose to 100 mg. Participants who had glasdegib dose reduction were reported as the starting glasdegib dose level received. Two (2) participants in this cohort had dose reduction to 100 mg starting from Cycle 2/Day 1 and Cycle 2/Day 16, respectively.
- Phase 1B: Glasdegib 100 mg + Decitabine: Participants received oral doses of glasdegib tablets 100 mg starting on Day 2 of Cycle 1 for PK assessment purposes and thereafter QD and continuously for 28-day cycles (starting on Day 1 for all other cycles). Decitabine was given at a dose of 20 mg/m^2 as an intravenous (IV) infusion over 1 hour on Days 1-5 of the 28-day cycles.
- Phase 1B: Glasdegib 200 mg + Decitabine: Participants received oral doses of glasdegib tablets 200 mg starting on Day 2 of Cycle 1 for PK assessment purposes and thereafter QD and continuously for 28-day cycles (starting on Day 1 for all other cycles). Decitabine was given at a dose of 20 mg/m^2 as an IV infusion over 1 hour on Days 1-5 of the 28-day cycles.In March 2013, all active participants receiving glasdegib 200 mg were required to reduce dose to 100 mg. Participants who had glasdegib dose reduction were reported as the starting glasdegib dose level received. Two (2) participants in this cohort had dose reduction to 100 mg starting from Cycle 1/Day 24 and Cycle 5/Day 1, respectively.
- Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin; Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin: Participants received 1-2 cycles of induction (glasdegib and daunorubicin/cytarabine), followed by 2-4 cycles of consolidation (glasdegib and high dose cytarabine) and a maximum of 6 cycles of maintenance (glasdegib alone). Daunorubicin was given on Days 1-3 QD at a dose of 60 mg/m^2/day by IV together with cytarabine on Days 1-7 at a dose of 100 mg/m^2/day by continuous IV infusion for each cycle of induction. Cytarabine was given on Days 1, 3, and 5 at a dose of 1 g/m^2 administered as a 3-hour IV infusion every 12 hours (2 g/m^2/day) for each cycle of consolidation. Glasdegib tablets 100 mg QD was started on induction Cycle 1/Day -3 and administered continuously QD thereafter for the duration of the study. A cycle was defined as 28 days.
- Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin: Participants received 1-2 cycles of induction (glasdegib and daunorubicin/cytarabine), followed by 2-4 cycles of consolidation (glasdegib and high dose cytarabine) and a maximum of 6 cycles of maintenance (glasdegib alone). Daunorubicin was given on Days 1-3 QD at a dose of 60 mg/m^2/day by IV together with cytarabine on Days 1-7 at a dose of 100 mg/m^2/day by continuous IV infusion for each cycle of induction. Cytarabine was given on Days 1, 3, and 5 at a dose of 1 g/m^2 administered as a 3-hour IV infusion every 12 hours (2 g/m^2/day) for each cycle of consolidation. Glasdegib tablets 200 mg QD was started on induction Cycle 1/Day -3 and administered continuously QD thereafter for the duration of the study. A cycle was defined as 28 days.In March 2013, all active participants receiving glasdegib 200 mg were required to reduce dose to 100 mg.One (1) participant in this cohort had dose reduction to 100 mg starting from Consolidation Cycle 1/Day 21.
- Phase 2 Unfit: Glasdegib 100 mg + LDAC: Participants received oral doses of glasdegib tablets 100 mg QD in 28-day cycles on a continuous basis, starting on Day 1 of Cycle 1. LDAC was given at a dose of 20 mg subcutaneously BID on Days 1-10 of the 28-day cycles.
- Phase 2 Unfit: LDAC Alone: Participants received LDAC subcutaneously at a dose of 20 mg BID on Days 1-10 of the 28-day cycles.
Period: Overall Study
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Started | 17 | 6 | 4 | 3 | 16 | 6 | 71 | 88 | 44
Received Treatment | 17 | 6 | 4 | 3 | 16 | 6 | 69 | 84 | 41
Completed | 1 | 0 | 0 | 0 | 6 | 2 | 18 | 4 | 1
Not Completed | 16 | 6 | 4 | 3 | 10 | 4 | 53 | 84 | 43
Not completed — Death | 15 | 6 | 4 | 2 | 9 | 3 | 46 | 76 | 39
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 3 | 1
Not completed — : Randomized, not treated | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Phase 1B: Glasdegib + LDAC: Included all participants who received oral glasdegib in combination with LDAC in phase 1B portion.
- Phase 1B: Glasdegib + Decitabine: Included all participants who received oral glasdegib in combination with decitabine in phase 1B portion.
- Phase 1B: Glasdegib + Cytarabine/Daunorubicin: Included all participants who received oral glasdegib in combination with cytarabine/daunorubicin in phase 1B portion.
- Total: Total of all reporting groups
Arm/Group | Phase 1B: Glasdegib + LDAC | Phase 1B: Glasdegib + Decitabine | Phase 1B: Glasdegib + Cytarabine/Daunorubicin | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone | Total
Number analyzed (Participants) | 23 | 7 | 22 | 71 | 88 | 44 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.8 (6.5) | 75.0 (4.4) | 54.9 (12.7) | 61.9 (9.6) | 76.2 (6.2) | 74.5 (4.9) | 66.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10 | 28 | 19 | 18 | 85
  Male | 15 | 5 | 12 | 43 | 69 | 26 | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) at Phase 1B
Description: A DLT was any of the following adverse events (AEs) in Cycle 1 and considered by the investigator possibly related to glasdegib in combination with chemotherapy: (1) Grade >= 3 non-hematologic toxicity, excluding Grade >= 3 infection, fever (including febrile neutropenia), infusion related AEs, electrolyte abnormalities and ALT/AST elevation that returned to Grade <= 1 or baseline within 7 days; (2) prolonged myelosuppression that lasted longer than 42 days from the point of detection, defined as absolute neutrophil count (ANC) < 500/microliter(mcL) or platelet count < 10 *10^9/L with a normal bone marrow (<5% blasts and no evidence of disease or dysplasia); (3) inability to deliver at least 80% of the planned study doses for all agents in a combination due to non-hematologic toxicities; (4) Delay of >28 days in receiving the next scheduled cycle due to persisting non-hematologic toxicities. Arm A: Glasdegib+LDAC; Arm B: Glasdegib+Decitabine; Arm C: Glasdegib+Cytarabine/Daunorubicin.
Time Frame: Arms A and B: Cycle 1, Day 1 to Day 28; Arm C: Cycle 1, Day -3 to Day 21 or to Day 28 depending on when the next chemotherapy cycle was started
Population: Per protocol analysis set: all enrolled participants in the dose escalation component who received at least 1 dose of glasdegib and of the co-administered chemotherapeutics and who did not have major treatment deviations during the DLT monitoring period.
Measure: Number; unit: Participants
Groups:
- Phase 1B: Glasdegib 100 mg + LDAC: Participants received oral doses of glasdegib (PF-04449913) tablets 100 milligram (mg) starting on Day 3 of Cycle 1 for pharmacokinetic (PK) assessment purposes and thereafter once daily (QD) and continuously for 28-day cycles (starting on Day 1 for all other cycles). LDAC was given at a dose of 20 mg subcutaneously twice daily (BID) on Days 1-10 of the 28-day cycles.
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 3 | 5 | 4 | 2 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Percentage of Participants With Complete Response (CR) at Phase 2 Fit
Description: For AML participants:CR were those with repeat bone marrow showing <5% myeloblasts,spicules present and no Auer rods, peripheral blood showing neutrophils>=1000/mcL and platelets>=100,000/mcL, transfusion independent and no extramedullary disease. For MDS participants:CR were those with repeat bone marrow showing <=5% myeloblasts, peripheral blood showing neutrophils>=1000/mcL, platelets>=100,000/mcL, 0% blast and hemoglobin (Hgb)>= 11 g/dL, normal maturation of all cell lines.
Time Frame: 4 years
Population: Full analysis set: all enrolled participants of Phase 2 Fit arm who received at least 1 dose of study medication. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 69
Percentage of participants
  Total participants | 42.0 [34.4 to 49.6]
  Participants >= 55 years old: number analyzed (Participants) | 60
  Participants >= 55 years old | 36.7 [28.7 to 44.6]
  Participants < 55 years old: number analyzed (Participants) | 9
  Participants < 55 years old | 77.8 [60.0 to 95.5]

3. Primary Outcome: Overall Survival (OS) at Phase 2 Unfit
Description: OS was defined as duration from the date of randomization to the date of death from any cause. Kaplan-Meier (KM) method was used to estimate median OS. In this method, every participant had a follow-up time which was associated with an indicator, 1=event (death in our case), and 0 =censored. If the participants were not known to have died, time to date of last known to be alive was used as to calculate the follow-up time and indicator was 0 for these participants. KM method estimates the median OS based on the K-M curve. The K-M curve only drops when we had an event and censor data are the ticks in the graph. To estimate median OS, the K-M curve usually will be smoothed first and a line will be drawn at 50%. The median OS is the point when K-M curve and the horizontal hit. Survival status was collected every month for the first 2 months after discontinuation of study treatment and thereafter every 2 months until death or 4 years from time of randomization for each participant.
Time Frame: Randomization to Follow-up (4 years)
Population: Full analysis set: all randomized participants of Phase 2 Unfit arm.
Measure: Median (80% Confidence Interval); unit: Months
Groups:
- Phase 2 Unfit: Glasdegib 100 mg + LDAC: Participants received oral doses of glasdegib tablets 100 mg QD in 28-day cycles on a continuous basis, starting on Day 1 of Cycle 1. LDAC was given at a dose of 20 mg subcutaneously BID on Days 1-10 of the 28 day cycles.
- Phase 2 Unfit: LDAC Alone: Participants received LDAC subcutaneously at a dose of 20 mg BID on Days 1-10 of the 28 day cycles.
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 88 | 44
Months | 8.8 [6.9 to 9.9] | 4.9 [3.5 to 6.0]
Statistical Analysis 1: Comparison: Phase 2 Unfit: Glasdegib 100 mg + LDAC vs Phase 2 Unfit: LDAC Alone; Test type: Other; p = 0.0020, Log Rank — 1-sided p-value from the log-rank test stratified by prognosis stratum according to Interactive Voice Response System (IVRS); Hazard Ratio (HR) = 0.569, 80% CI 2-sided [0.441 to 0.734] — Based on the Cox proportional hazards model stratified by prognosis stratum according to IVRS

4. Secondary Outcome: Overall Survival (OS) at Phase 1B
Description: OS was defined as duration from the date of randomization to the date of death from any cause. Kaplan-Meier (KM) method was used to estimate median OS. In this method, every participant had a follow-up time which was associated with an indicator, 1=event (death in our case), and 0 =censored. If the participants were not known to have died, time to date of last known to be alive was used as to calculate the follow-up time and indicator was 0 for these participants. KM method estimates the median OS based on the K-M curve. The K-M curve only drops when we had an event and censor data are the ticks in the graph. To estimate median OS, the K-M curve usually will be smoothed first and a line will be drawn at 50%. The median OS is the point when K-M curve and the horizontal hit. Survival status was collected every month for the first 2 months after discontinuation of study treatment and thereafter every 2 months until death or 4 years from each participant's first dose.
Time Frame: First dose to Follow-up (4 years)
Population: Full analysis set: all enrolled participants of Phase 1B portion who received at least 1 dose of study medication.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Phase 1B: Glasdegib + LDAC | Phase 1B: Glasdegib + Decitabine | Phase 1B: Glasdegib + Cytarabine/Daunorubicin
Number analyzed (Participants) | 23 | 7 | 22
Months | 4.4 [2.5 to 6.6] | 11.5 [4.5 to 17.4] | 37.8 [14.5 to NA] — The upper bound of 80% CI was not estimable, as 10 (45.5%) participants were censored for no longer being followed for survival

5. Secondary Outcome: Overall Survival (OS) at Phase 2 Fit
Description: as for outcome 4
Time Frame: First dose to Follow-up (4 years)
Population: as for outcome 2
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 69
Months
  Total participants | 14.9 [13.4 to 19.3]
  Participants >= 55 years old: number analyzed (Participants) | 60
  Participants >= 55 years old | 14.7 [13.1 to 17.7]
  Participants < 55 years old: number analyzed (Participants) | 9
  Participants < 55 years old | NA [11.0 to NA] — Number of deaths was 4 until the study completion, not enough for OS calculation.

6. Secondary Outcome: Percentage of Participants With CR / Complete Response With Incomplete Blood Count Recovery (CRi) at Phase 1B
Description: For AML participants:CR were those with repeat bone marrow showing <5% myeloblasts,spicules present and no Auer rods, peripheral blood showing neutrophils>=1000/mcL and platelets>=100,000/mcL, transfusion independent and no extramedullary disease. For MDS participants:CR were those with repeat bone marrow showing <=5% myeloblasts, peripheral blood showing neutrophils>=1000/mcL, platelets>=100,000/mcL, 0% blast and hemoglobin (Hgb)>= 11 g/dL, normal maturation of all cell lines.For AML and MDS participants, complete response with incomplete blood count recovery(CRi)were those with repeat bone marrow showing <5% myeloblasts with either platelets or neutrophils not recovered (platelets <100,000/mcL or neutrophils <1000/mcL).
Time Frame: 4 years
Population: Full analysis set: all enrolled participants of Phase 1B portion who received at least 1 dose of study medication.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1B: Glasdegib + LDAC | Phase 1B: Glasdegib + Decitabine | Phase 1B: Glasdegib + Cytarabine/Daunorubicin
Number analyzed (Participants) | 23 | 7 | 22
Percentage of participants | 8.7 [2.3 to 21.5] | 28.6 [7.9 to 59.6] | 54.5 [38.9 to 69.5]

7. Secondary Outcome: Percentage of Participants With Complete Response (CR) at Phase 2 Unfit
Description: as for outcome 2
Time Frame: 4 years
Population: Full analysis set: all randomized participants of Phase 2 Unfit arm.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 88 | 44
Percentage of participants | 18.2 [12.9 to 23.5] | 2.3 [0.0 to 5.2]
Statistical Analysis 1: Comparison: Phase 2 Unfit: Glasdegib 100 mg + LDAC vs Phase 2 Unfit: LDAC Alone; Test type: Other; p = 0.0112, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.2755, 80% CI 2-sided [1.3057 to 13.9994] — Based on the Cox proportional hazards model stratified by prognosis stratum according to IVRS

8. Secondary Outcome: Percentage of Participants With Disease-specific Efficacy for Acute Myeloid Leukemia (AML) at Phase 2 Fit and Unfit
Description: AML participants,disease specific efficacy measures included:CRi;Morphologic Leukemia Free State(MLFS)(bone marrow<5%myeloblasts with spicules and no blasts with auer rods,neutrophils<1000/mcL and platelets<100,000/mcL);partial remission(PR)(bone marrow myeloblasts decrease to 5-25&>=50%decrease from start, neutrophils>=1000/mcL, platelets>=100,000/mcL);PR with incomplete blood count recovery(PRi)(bone marrow myeloblasts decrease to 5-25&>=50%decrease from start,neutrophils<1000/mcL or platelets<100,000/mcL);minor response(MR)(bone marrow myeloblasts decrease to>=25% from start);stable disease(SD)(bone marrow myeloblasts stable+/-25% from screening value);cytogenetic complete response(CRc)(bone marrow<5%myeloblasts, neutrophils>1000/mcL, platelets>100,000/mcL and normal cytogenetics),molecular complete response(CRm)(bone marrow<5%myeloblasts, neutrophils>1000/mcL, platelets>100,000/mcL and molecular-negative).
Time Frame: 4 years
Population: AML participants in the Full analysis set: all enrolled participants of Phase 2 Fit arm who received at least 1 dose of study medication, and all randomized participants of Phase 2 Unfit arm.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 64 | 78 | 38
Percentage of participants
  CRi | 10.9 [6.2 to 17.7] | 5.1 [2.3 to 10.0] | 2.6 [0.3 to 9.9]
  MLFS | 7.8 [3.8 to 14.0] | 2.6 [0.7 to 6.7] | 0.0 [0.0 to 5.9]
  PR | 1.6 [0.2 to 5.9] | 6.4 [3.2 to 11.6] | 2.6 [0.3 to 9.9]
  PRi | 1.6 [0.2 to 5.9] | 1.3 [0.1 to 4.9] | 0.0 [0.0 to 5.9]
  MR | 10.9 [6.2 to 17.7] | 6.4 [3.2 to 11.6] | 10.5 [4.7 to 19.9]
  SD | 6.3 [2.8 to 12.1] | 16.7 [11.3 to 23.4] | 21.1 [12.7 to 31.9]
  CRc | 35.9 [27.9 to 44.7] | 11.5 [7.1 to 17.6] | 0.0 [0.0 to 5.9]
  CRm | 37.5 [29.4 to 46.2] | 16.7 [11.3 to 23.4] | 2.6 [0.3 to 9.9]

9. Secondary Outcome: Percentage of Participants With Disease-specific Efficacy for Myelodysplastic Syndrome (MDS) at Phase 2 Fit and Unfit
Description: For all MDS participants, disease specific efficacy measures included: CRi (bone marrow showing <5% myeloblasts with platelets <100,000/mcL or neutrophils <1000/mcL, including confirmed and unconfirmed responses); PR (repeat bone marrow myeloblasts showing decreased by >= 50% decrease but still >5%, peripheral blood showing neutrophils >= 1,000/mcL, platelets >= 100,000/mcL and Hgb>=11g/dL; including confirmed and unconfirmed responses); SD (including confirmed and unconfirmed responses, failure to achieve PR and no evidence of progression for >8 weeks); marrow complete response (mCR) (bone marrow showing <=5% myeloblasts and decreased by >= 50%), partial cytogenetic response (>=50% reduction of chromosomal abnormality) and complete cytogenetic response (CRc) (disappearance of chromosomal abnormality with no appearance of now ones).
Time Frame: 4 years
Population: MDS participants in the Full analysis set: all enrolled participants of Phase 2 Fit arm who received at least 1 dose of study medication, and all randomized participants of Phase 2 Unfit arm.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 5 | 10 | 6
Percentage of participants
  mCR | 0.0 [0.0 to 36.9] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 31.9]
  PR | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 31.9]
  SD | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 20.6] | 33.3 [9.3 to 66.7]
  CRi | 20.0 [2.1 to 58.4] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 31.9]
  Unconfirmed SD | 0.0 [0.0 to 36.9] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 31.9]
  Unconfirmed CRi | 0.0 [0.0 to 36.9] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 31.9]
  mCR (CRi not included) | 0.0 [0.0 to 36.9] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 31.9]
  CRc | 60.0 [24.7 to 88.8] | 10.0 [1.0 to 33.7] | 0.0 [0.0 to 31.9]

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Glasdegib in Participants Receiving Glasdegib and LDAC at Phase 1B on Cycle 1/Day 10 and Cycle 1/Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post-dose on Cycle 1/Day 10 and Cycle 1/Day 21
Population: Dose compliant group:Participants who had at least 4 days of uninterrupted dosing for a multiple dose PK assessment were considered to be at steady state,part of the "dose compliant" group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC
Number analyzed (Participants) | 17 | 6
ng/mL
  Cycle 1/Day 10: number analyzed (Participants) | 13 | 6
  Cycle 1/Day 10 | 1074 (63) | 1942 (75)
  Cycle 1/Day 21: number analyzed (Participants) | 8 | 5
  Cycle 1/Day 21 | 1242 (56) | 2577 (104)

11. Secondary Outcome: Time to Cmax (Tmax) of Glasdegib in Participants Receiving Glasdegib and LDAC at Phase 1B on Cycle 1/Day 10 and Cycle 1/Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post-dose on Cycle 1/Day 10 and Cycle 1/Day 21
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC
Number analyzed (Participants) | 17 | 6
Hours
  Cycle 1/Day 10: number analyzed (Participants) | 13 | 6
  Cycle 1/Day 10 | 1.75 [0.750 to 24.0] | 4.00 [1.02 to 24.0]
  Cycle 1/Day 21: number analyzed (Participants) | 8 | 5
  Cycle 1/Day 21 | 1.34 [0.533 to 2.00] | 4.00 [1.00 to 6.00]

12. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to Dosing Interval (AUCtau) of Glasdegib in Participants Receiving Glasdegib and LDAC at Phase 1B on Cycle 1/Day 10 and Cycle 1/Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post-dose on Cycle 1/Day 10 and Cycle 1/Day 21
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC
Number analyzed (Participants) | 17 | 6
ng*hr/mL
  Cycle 1/Day 10: number analyzed (Participants) | 10 | 4
  Cycle 1/Day 10 | 15020 (49) | 28600 (17)
  Cycle 1/Day 21: number analyzed (Participants) | 8 | 4
  Cycle 1/Day 21 | 16660 (43) | 31400 (119)

13. Secondary Outcome: Cmax of Glasdegib in Participants Receiving Glasdegib and Decitabine at Phase 1B on Cycle 1/Day 10 and Cycle 2/Day 1
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post-dose on Cycle 1/Day 10; pre-dose, 0.5, 1, 2, 6 and 24 hours post-dose on Cycle 2/Day 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine
Number analyzed (Participants) | 4 | 3
ng/mL
  Cycle 1/Day 10: number analyzed (Participants) | 3 | 3
  Cycle 1/Day 10 | 1718 (28) | 2381 (28)
  Cycle 2/Day 1: number analyzed (Participants) | 3 | 2
  Cycle 2/Day 1 | 1826 (44) | NA (NA) — Based on pre-specified criteria, statistical analysis was not performed if fewer than 3 participants have reportable parameter values.

14. Secondary Outcome: Tmax of Glasdegib in Participants Receiving Glasdegib and Decitabine at Phase 1B on Cycle 1/Day 10 and Cycle 2/Day 1
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine
Number analyzed (Participants) | 4 | 3
Hours
  Cycle 1/Day 10: number analyzed (Participants) | 3 | 3
  Cycle 1/Day 10 | 2.00 [0.500 to 24.0] | 2.05 [1.00 to 5.97]
  Cycle 2/Day 1: number analyzed (Participants) | 3 | 2
  Cycle 2/Day 1 | 1.03 [0.567 to 2.00] | NA [NA to NA] — Based on pre-specified criteria, statistical analysis was not performed if fewer than 3 participants have reportable parameter values.

15. Secondary Outcome: AUCtau of Glasdegib in Participants Receiving Glasdegib and Decitabine at Phase 1B on Cycle 1/Day 10 and Cycle 2/Day 1
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine
Number analyzed (Participants) | 4 | 3
ng*hr/mL
  Cycle 1/Day 10: number analyzed (Participants) | 2 | 3
  Cycle 1/Day 10 | NA (NA) — Based on pre-specified criteria, statistical analysis was not performed if fewer than 3 participants have reportable parameter values. Individual AUCtau values are 17700 and 26300 ng*hr/mL. | 28380 (11)
  Cycle 2/Day 1: number analyzed (Participants) | 3 | 2
  Cycle 2/Day 1 | 17060 (29) | NA (NA) — Based on pre-specified criteria, statistical analysis was not performed if fewer than 3 participants have reportable parameter values.

16. Secondary Outcome: Cmax of Glasdegib in Participants Receiving Glasdegib and Cytarabine/Daunorubicin at Phase 1B on Induction Cycle 1/Day 3 and Day 10
Time Frame: Pre-dose, 0.5, 1, 6 and 24 hours post-dose on Induction Cycle 1/Day 3; pre-dose, 0.5, 1, 4, 6 and 24 hours post-dose on Induction Cycle 1/Day 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 16 | 6
ng/mL
  Induction Cycle 1/Day 3: number analyzed (Participants) | 14 | 6
  Induction Cycle 1/Day 3 | 674.2 (45) | 1622 (25)
  Induction Cycle 1/Day 10: number analyzed (Participants) | 15 | 6
  Induction Cycle 1/Day 10 | 1135 (43) | 2371 (43)

17. Secondary Outcome: Tmax of Glasdegib in Participants Receiving Glasdegib and Cytarabine/Daunorubicin at Phase 1B on Induction Cycle 1/Day 3 and Day 10
Time Frame: as for outcome 16
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 16 | 6
Hours
  Induction Cycle 1/Day 3: number analyzed (Participants) | 14 | 6
  Induction Cycle 1/Day 3 | 5.99 [0.467 to 25.2] | 6.00 [1.00 to 6.07]
  Induction Cycle 1/Day 10: number analyzed (Participants) | 15 | 6
  Induction Cycle 1/Day 10 | 4.08 [0.500 to 24.7] | 1.04 [0.583 to 4.12]

18. Secondary Outcome: AUCtau of Glasdegib in Participants Receiving Glasdegib and Cytarabine/Daunorubicin at Phase 1B on Induction Cycle 1/Day 3 and Day 10
Time Frame: as for outcome 16
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 16 | 6
ng*hr/mL
  Induction Cycle 1/Day 3: number analyzed (Participants) | 12 | 5
  Induction Cycle 1/Day 3 | 9332 (56) | 22840 (43)
  Induction Cycle 1/Day 10: number analyzed (Participants) | 13 | 5
  Induction Cycle 1/Day 10 | 16300 (46) | 26370 (39)

19. Secondary Outcome: Cmax of LDAC and Ara-U in Participants Receiving Glasdegib and LDAC at Phase 1B on Cycle 1/Day 2 and Cycle 1/Day 10
Description: Ara-U is the major metabolite of cytarabine. LDAC (low dose cytarabine) is rapidly degraded to the stable metabolite Ara-U, Cmax levels of both LDAC and Ara-U were reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4 and 6 hours post-dose on Cycle 1/Day 2 and Cycle 1/Day 10
Population: PK concentration population: all treated participants who had at least 1 concentration of any of the study drugs.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC
Number analyzed (Participants) | 17 | 6
ng/mL
  LDAC Cycle 1/Day 2: number analyzed (Participants) | 16 | 6
  LDAC Cycle 1/Day 2 | 58.50 (58) | 100.1 (29)
  LDAC Cycle 1/Day 10: number analyzed (Participants) | 12 | 6
  LDAC Cycle 1/Day 10 | 63.01 (88) | 132.5 (39)
  Ara-U Cycle 1/Day 2 | 379.5 (34) | 569.7 (29)
  Ara-U Cycle 1/Day 10: number analyzed (Participants) | 12 | 6
  Ara-U Cycle 1/Day 10 | 452.2 (36) | 652.0 (27)

20. Secondary Outcome: Tmax of LDAC and Ara-U in Participants Receiving Glasdegib and LDAC at Phase 1B on Cycle 1/Day 2 and Cycle 1/Day 10
Description: Ara-U is the major metabolite of cytarabine. LDAC (low dose cytarabine) is rapidly degraded to the stable metabolite Ara-U, Tmax levels of both LDAC and Ara-U were reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4 and 6 hours post-dose on Cycle 1/Day 2 and Cycle 1/Day 10
Population: PK parameter analysis set: all treated participants who had at least 1 of the PK parameters of interest for any of the study drugs.
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC
Number analyzed (Participants) | 17 | 6
Hours
  LDAC Cycle 1/Day 2: number analyzed (Participants) | 16 | 6
  LDAC Cycle 1/Day 2 | 0.250 [0.233 to 1.00] | 0.250 [0.250 to 0.500]
  LDAC Cycle 1/Day 10: number analyzed (Participants) | 12 | 6
  LDAC Cycle 1/Day 10 | 0.325 [0.233 to 1.00] | 0.250 [0.233 to 0.500]
  Ara-U Cycle 1/Day 2 | 3.97 [1.00 to 6.05] | 4.00 [1.00 to 6.00]
  Ara-U Cycle 1/Day 10: number analyzed (Participants) | 12 | 6
  Ara-U Cycle 1/Day 10 | 2.00 [0.000 to 6.00] | 1.99 [1.02 to 4.08]

21. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to Infinity (AUCinf) of LDAC in Participants Receiving Glasdegib and LDAC at Phase 1B on Cycle 1/Day 2 and Cycle 1/Day 10
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4 and 6 hours post-dose on Cycle 1/Day 2 and Cycle 1/Day 10
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC
Number analyzed (Participants) | 17 | 6
ng*hr/mL
  LDAC Cycle 1/Day 2: number analyzed (Participants) | 14 | 6
  LDAC Cycle 1/Day 2 | 71.10 (28) | 89.35 (28)
  LDAC Cycle 1/Day 10: number analyzed (Participants) | 9 | 5
  LDAC Cycle 1/Day 10 | 92.28 (25) | 143.9 (24)

22. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of LDAC and Ara-U in Participants Receiving Glasdegib and LDAC at Phase 1B on Cycle 1/Day 2 and Cycle 1/Day 10
Description: Ara-U is the major metabolite of cytarabine. LDAC (low dose cytarabine) is rapidly degraded to the stable metabolite Ara-U. Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast) levels of both LDAC and Ara-U were reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4 and 6 hours post-dose on Cycle 1/Day 2 and Cycle 1/Day 10
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC
Number analyzed (Participants) | 17 | 6
ng*hr/mL
  LDAC Cycle 1/Day 2: number analyzed (Participants) | 16 | 6
  LDAC Cycle 1/Day 2 | 62.55 (41) | 87.49 (29)
  LDAC Cycle 1/Day 10: number analyzed (Participants) | 12 | 6
  LDAC Cycle 1/Day 10 | 65.56 (76) | 134.8 (26)
  Ara-U Cycle 1/Day 2 | 2036 (36) | 3050 (29)
  Ara-U Cycle 1/Day 10: number analyzed (Participants) | 12 | 6
  Ara-U Cycle 1/Day 10 | 2283 (43) | 3528 (29)

23. Secondary Outcome: Cmax of Decitabine in Participants Receiving Glasdegib and Decitabine at Phase 1B on Cycle 1/Day 1 and Cycle 1/Day 2
Time Frame: Pre-dose, 0.5 hour from start of infusion, 1 hour (at end of infusion) and 2, 3 and 4 hours from start of infusion on Cycle 1/Day 1 and Cycle 1/Day 2
Population: PK concentration population: all treated participants who had at least 1 concentration of any of the study drugs.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Phase 1B: Glasdegib 200 mg + Decitabine: Participants received oral doses of glasdegib tablets 200 mg starting on Day 3 of Cycle 1 for PK assessment purposes and thereafter QD and continuously for 28-day cycles (starting on Day 1 for all other cycles). LDAC was given at a dose of 20 mg subcutaneously BID on Days 1-10 of the 28-day cycles. In March 2013, all active participants receiving glasdegib 200 mg were required to reduce dose to 100 mg. Participants who had glasdegib dose reduction were reported as the starting glasdegib dose level received. Two (2) participants in this cohort had dose reduction to 100 mg starting from Cycle 2/Day 1 and Cycle 2/Day 16, respectively.
Arm/Group | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine
Number analyzed (Participants) | 4 | 3
ng/mL
  Cycle 1/Day 1: number analyzed (Participants) | 3 | 3
  Cycle 1/Day 1 | 113.4 (59) | 174.2 (113)
  Cycle 1/Day 2: number analyzed (Participants) | 3 | 3
  Cycle 1/Day 2 | 127.9 (43) | 121.7 (37)

24. Secondary Outcome: Tmax of Decitabine in Participants Receiving Glasdegib and Decitabine at Phase 1B on Cycle 1/Day 1 and Cycle 1/Day 2
Time Frame: as for outcome 23
Population: as for outcome 20
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine
Number analyzed (Participants) | 4 | 3
Hours
  Cycle 1/Day 1: number analyzed (Participants) | 3 | 3
  Cycle 1/Day 1 | 0.75 [0.50 to 1.0] | 0.53 [0.52 to 0.75]
  Cycle 1/Day 2: number analyzed (Participants) | 3 | 3
  Cycle 1/Day 2 | 0.58 [0.53 to 0.95] | 0.53 [0.52 to 1.3]

25. Secondary Outcome: AUCinf of Decitabine in Participants Receiving Glasdegib and Decitabine at Phase 1B on Cycle 1/Day 1 and Cycle 1/Day 2
Time Frame: as for outcome 23
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine
Number analyzed (Participants) | 4 | 3
ng*hr/mL
  Cycle 1/Day 1: number analyzed (Participants) | 3 | 3
  Cycle 1/Day 1 | 133.4 (71) | 251.5 (140)
  Cycle 1/Day 2: number analyzed (Participants) | 2 | 2
  Cycle 1/Day 2 | NA (NA) — Based on pre-specified criteria, statistical analysis was not performed if fewer than 3 participants have reportable parameter values. Individual AUCinf values are 265 and 1040 ng*hr/mL. | NA (NA) — Based on pre-specified criteria, statistical analysis was not performed if fewer than 3 participants have reportable parameter values. Individual AUCinf values are 154 and 216 ng*hr/mL.

26. Secondary Outcome: AUCtau of Cytarabine and Ara-U in Participants Receiving Glasdegib and Cytarabine/Daunorubicin at Phase 1B on Induction Cycle 1/Day 3
Description: Ara-U is the major metabolite of cytarabine. LDAC (low dose cytarabine) is rapidly degraded to the stable metabolite Ara-U, levels of both cytarabine and Ara-U were reported.
Time Frame: Pre-dose, 6 and 24 hours post start of cytarabine infusion on Induction Cycle 1/Day 3
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 9 | 2
ng*hr/mL
  Cytarabine | 1070 (211) | NA (NA) — Based on pre-specified criteria, statistical analysis was not performed if fewer than 3 participants have reportable parameter values. Individual AUCtau values are 276 and 879 ng*hr/mL.
  Ara-U | 28420 (32) | NA (NA) — Based on pre-specified criteria, statistical analysis was not performed if fewer than 3 participants have reportable parameter values. Individual AUCtau values are 32430 and 45900 ng*hr/mL.

27. Secondary Outcome: Cmax of Daunorubicin and Daunorubicinol in Participants Receiving Glasdegib and Cytarabine/Daunorubicin at Phase 1B on Induction Cycle 1/Day 3
Description: Daunorubicinol is the major metabolite of daunorubicin, which has anti-neoplastic activity. Cmax values of daunorubicin and daunorubicinol are reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 4, 6, 24 hours post administration of daunorubicin on Induction Cycle 1/Day 3
Population: PK concentration population: all treated participants who had at least 1 concentration of any of the study drugs.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 15 | 6
ng/mL
  Daunorubicin | 275.3 (153) | 341.0 (82)
  Daunorubicinol | 195.4 (139) | 233.4 (46)

28. Secondary Outcome: Tmax of Daunorubicin and Daunorubicinol in Participants Receiving Glasdegib and Cytarabine/Daunorubicin at Phase 1B on Induction Cycle 1/Day 3
Description: Daunorubicinol is the major metabolite of daunorubicin, which has anti-neoplastic activity. Tmax values of daunorubicin and daunorubicinol are reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 4, 6, 24 hours post administration of daunorubicin on Induction Cycle 1/Day 3
Population: as for outcome 20
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 15 | 6
Hours
  Daunorubicin | 0.500 [0.217 to 1.72] | 0.492 [0.250 to 0.600]
  Daunorubicinol | 1.00 [0.217 to 5.90] | 0.642 [0.283 to 4.00]

29. Secondary Outcome: AUCtau of Daunorubicin and Daunorubicinol in Participants Receiving Glasdegib and Cytarabine/Daunorubicin at Phase 1B on Induction Cycle 1/Day 3
Description: Daunorubicinol is the major metabolite of daunorubicin, which has anti-neoplastic activity. AUCtau values of daunorubicin and daunorubicinol are reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 4, 6, 24 hours post administration of daunorubicin on Induction Cycle 1/Day 3
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 16 | 6
ng*hr/mL
  Daunorubicin: number analyzed (Participants) | 14 | 4
  Daunorubicin | 499.3 (61) | 424.9 (38)
  Daunorubicinol: number analyzed (Participants) | 15 | 5
  Daunorubicinol | 2152 (24) | 2712 (33)

30. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of Glasdegib in Phase 2 Fit on Induction Cycle 1/Day 10
Time Frame: Pre-dose, 1 and 4 hours post-dose on Induction Cycle 1/Day 10
Population: Dose compliant, non CYP3A4 group: dose compliant group participants who did not have administration of any strong or moderate CYP3A4 inhibitors.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 42
ng/mL | 308.7 (74)

31. Secondary Outcome: Cmax of Glasdegib in Participants Receiving Glasdegib and LDAC at Phase 2 Unfit on Cycle 1/Day 10
Time Frame: Pre-dose, 1, 2, 4, and 6 hour post-dose on Cycle 1/Day 10
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC
Number analyzed (Participants) | 41
ng/mL | 1252 (44) [0.667 to 5.83]

32. Secondary Outcome: Tmax of Glasdegib in Participants Receiving Glasdegib and LDAC at Phase 2 Unfit on Cycle 1/Day 10
Time Frame: Pre-dose, 1, 2, 4, and 6 hour post-dose on Cycle 1/Day 10
Population: as for outcome 30
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC
Number analyzed (Participants) | 41
Hours | 1.67 [0.667 to 5.83]

33. Secondary Outcome: AUCtau of Glasdegib in Participants Receiving Glasdegib and LDAC at Phase 2 Unfit on Cycle 1/Day 10
Time Frame: Pre-dose, 1, 2, 4, and 6 hour post-dose on Cycle 1/Day 10
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC
Number analyzed (Participants) | 37
ng*hr/mL | 17210 (54) [0.667 to 5.83]

34. Secondary Outcome: Number of Participants With Disease-related Gene Mutations at Phase 1B
Description: Peripheral blood and bone marrow aspirate were collected for baseline mutational analyses. Genetic abnormalities frequently associated with AML were analyzed. These genetic abnormalities included known mutations in the genes NPM1, CEBPA, FLT3, RUNX1, IDH1, IDH2, KIT, K Ras, N Ras and WT1. Additional genes with mutations known to be associated with AML and MDS such as TET2 and DNMT3A were also evaluated.
Time Frame: Baseline (Cycle 1/Day 1 pre-dose for Glasdegib + LDAC and Glasdegib + Decitabine Arms; Induction Cycle 1/Day -3 pre-dose for Glasdegib +Cytarabine/Daunorubicin Arm)
Population: Pharmacodynamic (PD) analysis set: all enrolled participants in the Phase 1B portion who received at least 1 dose of glasdegib; responders and non-responders in each arm with at least 1 PD parameter from the corresponding assay sample with a baseline and an adequate post treatment assessment.
Measure: Number; unit: Participants
Groups:
- Phase 1B: Glasdegib + LDAC (Biomarker, Responder); Phase 1B: Glasdegib + Decitabine (Biomarker,Responder): AML participants who achieved CR, CRi, MLFS, PR, or PRi (AML investigator reported best overall response), and MDS participants who achieved CR, mCR, PR, or SD (MDS investigator reported best overall response).
- Phase 1B: Glasdegib + LDAC (Biomarker, Non-Responder): AML subjects who did not achieve CR, CRi, MLFS, PR, or PRi; and MDS subjects who did not achieve CR, mCR, PR or SD were defined as non-responders for best overall response.
- Phase 1B: Glasdegib + Decitabine (Biomaker,Non-Responder): AML participants who did not achieve CR, CRi, MLFS, PR, or PRi; and MDS participants who did not achieve CR, mCR, PR or SD were defined as non-responders for best overall response.
- Phase 1B: Glasdegib + Cytarabine/Dauno (Biomarker, Responder): AML subjects who achieved CR, CRi, MLFS, PR, or PRi (AML investigator reported best overall response), and MDS subjects who achieved CR, mCR, PR, or SD (MDS investigator reported best overall response). Dauno is short for daunorubicin.
- Phase 1B: Glasdegib+Cytarabine/Dauno(Biomarker,Non-Responder): AML participants who did not achieve CR, CRi, MLFS, PR, or PRi; and MDS participants who did not achieve CR, mCR, PR or SD were defined as non-responders for best overall response. Dauno is short for daunorubicin.
Arm/Group | Phase 1B: Glasdegib + LDAC (Biomarker, Responder) | Phase 1B: Glasdegib + LDAC (Biomarker, Non-Responder) | Phase 1B: Glasdegib + Decitabine (Biomarker,Responder) | Phase 1B: Glasdegib + Decitabine (Biomaker,Non-Responder) | Phase 1B: Glasdegib + Cytarabine/Dauno (Biomarker, Responder) | Phase 1B: Glasdegib+Cytarabine/Dauno(Biomarker,Non-Responder)
Number analyzed (Participants) | 0 | 9 | 0 | 1 | 11 | 1
Participants
  CEBPA (CCAAT/enhancer-binding protein alpha) |  | 3 |  | 0 | 2 | 0
  DNMT3A (DNA [cytosine-5]-methyltransferase 3A) |  | 2 |  | 0 | 0 | 0
  FLT3 (Fms-like tyrosine kinase 3) |  | 1 |  | 0 | 2 | 0
  FLT3-ITD (FLT3 internal tandem duplications) |  | 0 |  | 0 | 1 | 0
  IDH1 (Isocitrate dehydrogenase 1) |  | 1 |  | 0 | 0 | 0
  IDH2 (Isocitrate dehydrogenase 2) |  | 0 |  | 0 | 2 | 0
  KIT(Tyrosine-protein kinase Kit) |  | 0 |  | 1 | 0 | 0
  KRAS(Kirsten rat sarcoma 2 viral oncogene homolog) |  | 1 |  | 0 | 0 | 0
  NPM1 (Nucleophosmin) |  | 0 |  | 0 | 4 | 0
  NRAS(Neuroblastoma RAS viral oncogene homolog) |  | 5 |  | 0 | 1 | 0
  RUNX1 (Runt related transcription factor 1) |  | 1 |  | 0 | 1 | 0
  TET2 (Tet methylcytosine dioxygenase 2) |  | 3 |  | 0 | 1 | 0
  WT1 (Wilm's tumour tumor suppressor gene1) |  | 0 |  | 0 | 0 | 0

35. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 1B - Baseline
Description: Serum levels were determined for 38 circulating proteins. Values showing statistically significant, ≥2-fold difference compared with baseline are reported here.
Time Frame: Baseline (Induction Cycle 1/Day -3 pre-dose)
Population: Pharmacodynamic (PD) analysis set: all enrolled participants in the Phase 1B portion who received at least 1 dose of glasdegib, and had at least 1 PD parameter from the corresponding assay sample with a baseline and an adequate post treatment assessment.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1B: Glasdegib + Cytarabine/Daunorubicin
Number analyzed (Participants) | 22
pg/mL
  MMP-3 (Matrix metalloproteinase-3) | 10200 [1700 to 44000]
  IL-8 (Interleukin-8) | 10.7 [0.00 to 71.00]
  BDNF (Brain-derived neurotrophic factor) | 1200 [0.00 to 22000]
  IL-5 (Interleukin-5) | 0.00 [0.00 to 0.00]
  VEGF (Vascular endothelial growth factor) | 88.00 [32.00 to 2000.00]
  MCP-1 (Monocyte chemotactic protein-1) | 180.5 [0.00 to 1850.00]
  ITAC:Interferon-inducible T-cell α chemoattractant | 0.00 [0.00 to 1900.00]

36. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 1B - Induction Cycle 1/Day 3
Description: Serum levels were determined for 38 circulating proteins. Values showing statistically significant, ≥2-fold difference compared with baseline are reported here. Statistically significant, >=2-fold baseline difference was only seen for MMP-3 (Matrix metalloproteinase-3) at Induction Cycle 1/Day 3.
Time Frame: Induction Cycle 1/Day 3, 1 Hour Post dose
Population: as for outcome 35
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1B: Glasdegib + Cytarabine/Daunorubicin
Number analyzed (Participants) | 21
pg/mL | 20000 [1600 to 111000]

37. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 1B - Induction Cycle 1/Day 10
Description: as for outcome 35
Time Frame: Induction Cycle 1/Day 10, 1 Hour Post dose
Population: PD analysis set: all enrolled participants in the Phase 1B portion who received at least 1 dose of glasdegib, and had at least 1 PD parameter from the corresponding assay sample with a baseline and an adequate post treatment assessment.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1B: Glasdegib + Cytarabine/Daunorubicin
Number analyzed (Participants) | 21
pg/mL
  IL-8 | 37.00 [7.90 to 128.00]
  BDNF | 200 [0.00 to 2800]
  IL-5 | 99.00 [0.00 to 2440.00]
  VEGF | 51.00 [0.00 to 149.00]
  MCP-1 | 684.00 [368.00 to 9780.00]
  ITAC | 0.00 [0.00 to 218.00]

38. Secondary Outcome: Baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 1B
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. A total of 38 proteins were analyzed. The data of analytes for which the serum level showed statistically significant correlation with clinical response in Arm C are reported. Baseline levels statistically associated with best overall response was only seen in SDF-1 (stromal cell-derived factor 1) in glasdegib+cytarabine/daunorubicin arm.
Time Frame: as for outcome 34
Population: as for outcome 37
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1B: Glasdegib + Cytarabine/Dauno (Biomarker, Responder) | Phase 1B: Glasdegib+Cytarabine/Dauno(Biomarker,Non-Responder)
Number analyzed (Participants) | 14 | 8
pg/mL | 2275.00 [1600.00 to 3700.00] | 3275.00 [1950.00 to 4730.00]

39. Secondary Outcome: Post-baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 1B - Induction Cycle 1/Lead-In
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. A total of 38 proteins were analyzed. The data of analytes for which the serum level showed statistically significant correlation with clinical response are reported. Post-baseline levels statistically significant associated with best overall response was only seen for MMP-3 (Matrix metalloproteinase-3) at Induction Cycle 1/Lead-in.
Time Frame: Induction Cycle 1/Lead-in, 1 Hour Post dose
Population: as for outcome 37
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase 1B: Glasdegib + Cytarabine/Dauno (Biomarker, Responder) | Phase 1B: Glasdegib+Cytarabine/Dauno(Biomarker,Non-Responder)
Number analyzed (Participants) | 14 | 8
ng/mL | 8.90 [2.20 to 51.00] | 10.50 [6.50 to 19.00]

40. Secondary Outcome: Post-baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 1B - Induction Cycle 1/Day 3
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. A total of 38 proteins were analyzed. The data of analytes for which the serum level showed statistically significant correlation with clinical response are reported. Post-baseline levels statistically significant associated with best overall response was only seen for SDF-1 (Stromal cell-derived factor 1) at Induction Cycle 1/Day 3.
Time Frame: Induction Cycle 1/Day 3, 1 Hour Post dose
Population: as for outcome 37
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1B: Glasdegib + Cytarabine/Dauno (Biomarker, Responder) | Phase 1B: Glasdegib+Cytarabine/Dauno(Biomarker,Non-Responder)
Number analyzed (Participants) | 13 | 8
pg/mL | 2510.00 [1530.00 to 3520.00] | 3260.00 [1350.00 to 4430.00]

41. Secondary Outcome: Number of Participants With Disease-related Gene Mutations at Phase 2 Fit and Unfit
Description: as for outcome 34
Time Frame: Baseline (Induction Cycle 1/Day -3 pre-dose for Phase 2 Fit; Cycle 1/Day 1 pre-dose for Phase 2 Unfit)
Population: PD analysis set: all enrolled participants in the Phase 2 Fit and Unfit portion who received at least 1 dose of glasdegib; responders and non-responders in each arm with at least 1 PD parameter from the corresponding assay sample with a baseline and an adequate post treatment assessment.
Measure: Number; unit: Participants
Groups:
- Phase 2 Fit (Biomarker, Responder): AML participants who achieved CR, CRi, MLFS, PR, or PRi (AML investigator reported best overall response), and MDS participants who achieved CR, mCR, PR, or SD (MDS investigator reported best overall response).
- Phase 2 Fit (Biomarker,Non-Responder): AML participants who did not achieve CR, CRi, MLFS, PR, or PRi; and MDS participants who did not achieve CR, mCR, PR or SD were defined as non-responders for best overall response.
- Phase 2 Unfit: Glasdegib 100 mg + LDAC (Biomarker, Responder); Phase 2 Unfit: LDAC Alone (Biomarker, Responder): AML subjects who achieved CR, CRi, MLFS, PR, or PRi (AML investigator reported best overall response), and MDS subjects who achieved CR, mCR, PR, or SD (MDS investigator reported best overall response).
- Phase 2 Unfit: Glasdegib 100 mg+LDAC(Biomarker, Non-Responder); Phase 2 Unfit: LDAC Alone (Biomarker, Non-Responder): AML subjects who did not achieve CR, CRi, MLFS, PR, or PRi; and MDS subjects who did not achieve CR, mCR, PR or SD were defined as non-responders for best overall response.
Arm/Group | Phase 2 Fit (Biomarker, Responder) | Phase 2 Fit (Biomarker,Non-Responder) | Phase 2 Unfit: Glasdegib 100 mg + LDAC (Biomarker, Responder) | Phase 2 Unfit: Glasdegib 100 mg+LDAC(Biomarker, Non-Responder) | Phase 2 Unfit: LDAC Alone (Biomarker, Responder) | Phase 2 Unfit: LDAC Alone (Biomarker, Non-Responder)
Number analyzed (Participants) | 32 | 18 | 21 | 40 | 1 | 26
Participants
  CEBPA | 6 | 3 | 3 | 5 | 0 | 3
  DNMT3A | 12 | 6 | 2 | 13 | 0 | 6
  FLT3 | 3 | 2 | 1 | 4 | 0 | 0
  FLT3-ITD | 2 | 1 | 1 | 2 | 0 | 2
  IDH1 | 2 | 1 | 5 | 5 | 0 | 2
  IDH2 | 5 | 4 | 2 | 10 | 0 | 5
  KIT | 2 | 1 | 1 | 2 | 0 | 1
  KRAS | 0 | 1 | 0 | 2 | 0 | 2
  NPM1 | 12 | 3 | 2 | 3 | 0 | 1
  NRAS | 5 | 1 | 1 | 4 | 0 | 3
  RUNX1 | 7 | 7 | 10 | 18 | 0 | 7
  TET2 | 7 | 5 | 7 | 8 | 1 | 8
  WT1 | 0 | 1 | 1 | 2 | 0 | 1

42. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 2 Fit - Induction Cycle 1/Day 3
Description: Serum levels were determined for 38 circulating proteins. Selected values showing statistically significant difference compared with baseline are reported here.
Time Frame: Induction Cycle 1/Day 3, 1 Hour Post dose
Population: PD analysis set: all enrolled participants in the Phase 2 Fit portion who received at least 1 dose of glasdegib, and had at least 1 PD parameter from the corresponding assay sample with a baseline and an adequate post treatment assessment.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 57
pg/mL
  Factor VII(activated blood coagulation factor VII) | 318000 [56000 to 620000]
  BDNF | 700 [0 to 6200]
  MMP-3 | 21000 [1700 to 107000]
  IL-8 | 28.00 [0.00 to 139.00]
  ITAC | 14.00 [0.00 to 535.00]

43. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 2 Fit - Induction Cycle 1/Day 10
Description: as for outcome 42
Time Frame: Induction Cycle 1/Day 10, 1 Hour Post dose
Population: as for outcome 42
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 62
pg/mL
  IL-1β (Interleukin-1β) | 8.50 [0.00 to 15.00]
  IL-6 | 17.00 [0.00 to 7320.00]
  Factor VII | 292500 [45000 to 641000]
  BDNF | 300 [0 to 15000]
  VEGF | 69.00 [0.00 to 140.00]
  MCP-1 | 594.00 [126.00 to 21200.00]
  MMP-3 | 12000 [3000 to 93000]
  IL-8 | 55.00 [0.00 to 8930.00]
  IL-5 | 85.00 [0.00 to 2240.00]
  ITAC | 0.00 [0.00 to 46.00]

44. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 2 Fit - Consolidation Cycle 1/Day 1
Description: as for outcome 42
Time Frame: Consolidation Cycle 1/Day 1, 1 Hour Post dose
Population: as for outcome 42
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 24
pg/mL
  MIP-1β (Macrophage Inflammatory Protein-1β) | 226.00 [0.00 to 6160.00]
  BDNF | 7000 [370 to 38000]
  VEGF | 232.50 [41.00 to 834.00]
  IL-8 | 9.90 [0.00 to 514.00]
  ITAC | 41.50 [10.00 to 117.00]

45. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 2 Fit - Consolidation Cycle 1/Day 10
Description: as for outcome 42
Time Frame: Consolidation Cycle 1/Day 10, Pre-dose
Population: as for outcome 42
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 20
pg/mL
  MIP-1β | 239.50 [0.00 to 6560.00]
  MCP-1 | 581.00 [192.00 to 3880.00]
  MMP-3 | 12000 [2700 to 48000]
  IL-8 | 11.00 [0.00 to 74.00]
  ITAC | 4.10 [0.00 to 27.00]

46. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 2 Fit - End of Treatment
Description: as for outcome 42
Time Frame: End of Treatment (maximum of 12 cycles from start of therapy or until disease progression or relapse, participant refusal or unacceptable toxicity occurred, whichever came first, an average of 1 year)
Population: as for outcome 42
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 42
pg/mL
  MIP-1β | 338.00 [0.00 to 4480.00]
  VEGF | 133.00 [0.00 to 2880.00]
  MCP-1 | 277.00 [0.00 to 7450.00]

47. Secondary Outcome: Baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 2 Fit
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. A total of 38 proteins were analyzed. Selected data of analyte for which the serum level showed statistically significant correlation with clinical response are reported.
Time Frame: Baseline (Induction Cycle 1/Day -3 pre-dose)
Population: as for outcome 42
Measure: Median (Full Range); unit: pg/mL
Groups:
- Phase 2 Fit (Biomarker, Responder): AML subjects who achieved CR, CRi, MLFS, PR, or PRi (AML investigator reported best overall response), and MDS subjects who achieved CR, mCR, PR, or SD (MDS investigator reported best overall response).
- Phase 2 Fit (Biomarker, Non-Responder): AML subjects who did not achieve CR, CRi, MLFS, PR, or PRi; and MDS subjects who did not achieve CR, mCR, PR or SD were defined as non-responders for best overall response.
Arm/Group | Phase 2 Fit (Biomarker, Responder) | Phase 2 Fit (Biomarker, Non-Responder)
Number analyzed (Participants) | 43 | 22
pg/mL | 323.00 [158.00 to 419.00] | 362.00 [225.00 to 758.00]

48. Secondary Outcome: Post-baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 2 Fit - Induction Cycle 1/Day 3
Description: as for outcome 47
Time Frame: Induction Cycle 1/Day 3, 1 Hour Post dose
Population: as for outcome 42
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Phase 2 Fit (Biomarker, Responder) | Phase 2 Fit (Biomarker, Non-Responder)
Number analyzed (Participants) | 37 | 20
pg/mL | 3.20 [0.00 to 26.00] | 10.90 [0.00 to 63.00]

49. Secondary Outcome: Post-baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 2 Fit - Induction Cycle 1/Day 10
Description: as for outcome 47
Time Frame: Induction Cycle 1/Day 10, 1 Hour Post dose
Population: as for outcome 42
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Phase 2 Fit (Biomarker, Responder) | Phase 2 Fit (Biomarker, Non-Responder)
Number analyzed (Participants) | 42 | 20
pg/mL | 1.20 [0.00 to 18.00] | 6.60 [0.00 to 88.00]

50. Secondary Outcome: Post-baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 2 Fit - End of Treatment
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. A total of 38 proteins were analyzed. Selected data of analytes for which the serum level showed statistically significant correlation with clinical response are reported.
Time Frame: as for outcome 46
Population: as for outcome 42
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Fit (Biomarker, Responder) | Phase 2 Fit (Biomarker, Non-Responder)
Number analyzed (Participants) | 27 | 15
pg/mL
  IL-1β | 9.70 [0.00 to 20.00] | 6.70 [0.00 to 20.00]
  IL-15 (Interleukin-15) | 700 [0 to 1300] | 600 [0 to 850]

51. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 2 Unfit - Cycle 1/Day 1
Description: Serum levels were determined for 38 circulating proteins. Selected value showing statistically significant difference compared with baseline is reported here.
Time Frame: Cycle 1/Day 1, 1 Hour Post dose
Population: PD analysis set: all enrolled participants in the Phase 2 Unfit portion who received at least 1 dose of glasdegib, and had at least 1 PD parameter from the corresponding assay sample with a baseline and an adequate post treatment assessment.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC
Number analyzed (Participants) | 18
pg/mL | 483.00 [40.00 to 1230.00]

52. Secondary Outcome: Serum Levels of Circulating Protein Analytes at Phase 2 Unfit - Cycle 1/Day 10
Description: Serum levels were determined for 38 circulating proteins. Selected values showing statistically significant differences compared with baseline are reported here. ITAC (Interferon-inducible T-cell α chemoattractant) level in LDAC alone arm at Cycle 1/Day 10 exhibited non-significant change from baseline but similar trends as in Glasdegib 100 mg+LDAC arm.
Time Frame: Cycle 1/Day 10, Pre-dose
Population: as for outcome 51
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 66 | 24
pg/mL
  BDNF | 500 [0 to 7200] | 200 [0 to 5100]
  ITAC | 7.5 [0.00 to 226.00] | 0.00 [0.00 to 71.00]

53. Secondary Outcome: Baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 2 Unfit
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. A total of 38 proteins were analyzed. The data of analytes for which the serum level showed statistically significant correlation with clinical response are reported.
Time Frame: Baseline (Cycle 1/Day 1 pre-dose)
Population: as for outcome 51
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC (Biomarker, Responder) | Phase 2 Unfit: Glasdegib 100 mg+LDAC(Biomarker, Non-Responder)
Number analyzed (Participants) | 28 | 44
pg/mL
  BDNF | 2000 [170 to 22000] | 900 [0 to 12000]
  ICAM-1 (Intercellular cell adhesion molecule-1) | 128000 [37000 to 287000] | 161000 [82000 to 580000]
  6CKINE | 223.50 [53.00 to 679.00] | 318.00 [128.00 to 911.00]
  BAFF (B-cell activating factor) | 704.50 [116.00 to 3000.00] | 1295.00 [199.00 to 6190.00]
  MIP-3β | 275.00 [86.00 to 2060.00] | 414.50 [109.00 to 2130.00]
  Eotaxin-1 (C-C motif chemokine 11) | 169.00 [0.00 to 333.00] | 0.00 [0.00 to 260.00]

54. Secondary Outcome: Post-baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 2 Unfit - Cycle 1/Day 1
Description: as for outcome 50
Time Frame: Cycle 1/Day 1, 1 Hour Post-dose
Population: as for outcome 51
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC (Biomarker, Responder) | Phase 2 Unfit: Glasdegib 100 mg+LDAC(Biomarker, Non-Responder)
Number analyzed (Participants) | 6 | 12
pg/mL
  Factor VII:activated blood coagulation factor VII | 311500 [48000 to 661000] | 234500 [147000 to 676000]
  IL-6 (Interleukin-6) | 0.00 [0.00 to 3.50] | 6.80 [0.00 to 62.00]

55. Secondary Outcome: Post-baseline Levels of Serum Circulating Protein Analytes Associated With Best Overall Response at Phase 2 Unfit - End of Treatment
Description: as for outcome 47
Time Frame: as for outcome 46
Population: as for outcome 51
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC (Biomarker, Responder) | Phase 2 Unfit: Glasdegib 100 mg+LDAC(Biomarker, Non-Responder)
Number analyzed (Participants) | 17 | 18
pg/mL | 0.00 [0.00 to 45.00] | 9.40 [0.00 to 52.00]

56. Secondary Outcome: Ratios of mRNA Levels to Baseline at Phase 2 Fit - Induction Cycle 1/Day 3
Description: Whole blood mRNA analyses were performed on 21 mRNA candidates. Values showing statistically significant, ≥2-fold differences compared with baseline are reported here. CDKN1A: cyclin-dependent kinase inhibitor 1A; SMO: mRNA encoding the glasdegib target Smoothened; PTCH2: Patched 2; MYCN: Neuroblastoma Myc oncogene.
Time Frame: Baseline (Induction Cycle 1/Day -3 pre-dose); Induction Cycle 1/Day 3, 1 Hour Post dose
Population: PD analysis set: all enrolled participants in Phase 2 Fit who received at least 1 dose of glasdegib, had at least 1 PD parameter with a baseline and an adequate post treatment assessment.
Measure: Median (Full Range); unit: ratio
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 62
ratio
  CDKN1A: number analyzed (Participants) | 54
  CDKN1A | 2.40 [0.08 to 53.17]
  SMO: number analyzed (Participants) | 18
  SMO | 4.80 [0.06 to 51.22]
  PTCH2: number analyzed (Participants) | 10
  PTCH2 | 0.60 [0.03 to 2.66]
  MYCN: number analyzed (Participants) | 38
  MYCN | 0.20 [0.00 to 248.53]

57. Secondary Outcome: Ratios of mRNA Levels to Baseline at Phase 2 Fit - End of Treatment
Description: Whole blood mRNA analyses were performed on 21 mRNA candidates. Selected values showing statistically significant differences compared with baseline are reported here. CCND2:G1/S-Specific Cyclin D2; MSI2: Musashi RNA Binding Protein 2; PTCH2: Patched 2.
Time Frame: Baseline (Induction Cycle 1/Day -3 pre-dose); End of Treatment (maximum of 12 cycles from start of therapy or until disease progression or relapse, participant refusal or unacceptable toxicity occurred, whichever came first, an average of 1 year)
Population: as for outcome 56
Measure: Median (Full Range); unit: ratio
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 62
ratio
  CCND2: number analyzed (Participants) | 42
  CCND2 | 0.80 [0.23 to 3.23]
  MSI2: number analyzed (Participants) | 42
  MSI2 | 0.80 [0.31 to 4.58]
  PTCH2: number analyzed (Participants) | 12
  PTCH2 | 0.70 [0.29 to 1.90]

58. Secondary Outcome: Ratios of mRNA Levels to Baseline at Phase 2 Unfit - End of Treatment
Description: Whole blood mRNA analyses were performed on 21 mRNA candidates. Only the analytes showing statistically significant change from baseline are reported here.
Time Frame: Baseline (Cycle 1/Day 1 pre-dose); End of Treatment (maximum of 12 cycles from start of therapy or until disease progression or relapse, participant refusal or unacceptable toxicity occurred, whichever came first, an average of 1 year)
Population: PD analysis set:all enrolled participants in Phase 2 Unfit who received at least 1 dose of glasdegib, had at least 1 PD parameter with a baseline and an adequate post treatment assessment.
Measure: Median (Full Range); unit: ratio
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC
Number analyzed (Participants) | 47
ratio
  CCND2: number analyzed (Participants) | 30
  CCND2 | 0.70 [0.06 to 2.35]
  SMO: number analyzed (Participants) | 20
  SMO | 0.40 [0.09 to 8.09]
  CCND1: number analyzed (Participants) | 17
  CCND1 | 0.40 [0.10 to 13.33]

59. Secondary Outcome: Baseline mRNA Levels Associated With Best Overall Response at Phase 2 Fit
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. Whole blood mRNA analyses were performed on 21 mRNA candidates. Baseline mRNA level showing statistically significant correlation with clinical response are reported. Baseline mRNA levels statistically significant associated with best overall response was only seen for CCND2 (G1/S-Specific Cyclin D2).
Time Frame: Baseline (Induction Cycle 1/Day -3 pre-dose)
Population: as for outcome 42
Measure: Median (Full Range); unit: Normalized expression units
Arm/Group | Phase 2 Fit (Biomarker, Responder) | Phase 2 Fit (Biomarker, Non-Responder)
Number analyzed (Participants) | 39 | 22
Normalized expression units | 10.9 [1.61 to 25.26] | 14.80 [5.03 to 23.74]

60. Secondary Outcome: Baseline mRNA Levels Associated With Best Overall Response at Phase 2 Unfit
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. Whole blood mRNA analyses were performed on 21 mRNA candidates. Baseline mRNA level showing statistically significant correlation with clinical response are reported. FOXM1: Forkhead box M1; PTCH1: Patched 1.
Time Frame: Baseline (Cycle 1/Day 1 pre-dose)
Population: as for outcome 58
Measure: Median (Full Range); unit: Normalized expression units
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC (Biomarker, Responder) | Phase 2 Unfit: Glasdegib 100 mg+LDAC(Biomarker, Non-Responder)
Number analyzed (Participants) | 33 | 55
Normalized expression units
  FOXM1: number analyzed (Participants) | 15 | 28
  FOXM1 | 0.20 [0.05 to 0.77] | 0.40 [0.09 to 1.86]
  PTCH1: number analyzed (Participants) | 14 | 27
  PTCH1 | 0.20 [0.07 to 0.58] | 0.10 [0.01 to 0.42]

61. Secondary Outcome: Ratios of mRNA Levels to Baseline Associated With Best Overall Response at Phase 2 Fit
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. Whole blood mRNA analyses were performed on 21 mRNA candidates. Ratios of mRNA level to baseline showing statistically significant correlation with clinical response are reported.
Time Frame: as for outcome 57
Population: as for outcome 56
Measure: Median (Full Range); unit: ratio
Arm/Group | Phase 2 Fit (Biomarker, Responder) | Phase 2 Fit (Biomarker, Non-Responder)
Number analyzed (Participants) | 45 | 26
ratio
  CCNE1: number analyzed (Participants) | 26 | 13
  CCNE1 | 0.60 [0.21 to 1.65] | 1.10 [0.28 to 3.82]
  MSI2: number analyzed (Participants) | 28 | 14
  MSI2 | 0.90 [0.31 to 4.58] | 0.50 [0.33 to 1.86]

62. Secondary Outcome: Ratios of mRNA Levels Associated With Best Overall Response at Phase 2 Unfit
Description: Responders were AML participants who achieved CR, CRi, MLFS, PR or PRi based on investigator-reported best overall response and MDS participants who achieved CR, mCR, PR or SD based on investigator-reported best overall response. Whole blood mRNA analyses were performed on 21 mRNA candidates. Ratios of mRNA level to baseline showing statistically significant correlation with clinical response are reported. Ratios of mRNA levels to baseline statistically significant associated with best overall response was only seen for MYCN (Neuroblastoma Myc oncogene) at Cycle 1/Day 1.
Time Frame: Baseline (Cycle 1/Day 1 pre-dose); Cycle 1/Day 1, 1 Hour Post dose
Population: as for outcome 51
Measure: Median (Full Range); unit: ratio
Groups:
- Phase 2 Unfit: Glasdegib 100 mg + LDAC (Biomarker, Responder): AML participants who achieved CR, CRi, MLFS, PR, or PRi (AML investigator reported best overall response), and MDS participants who achieved CR, mCR, PR, or SD (MDS investigator reported best overall response).
Arm/Group | Phase 2 Unfit: Glasdegib 100 mg + LDAC (Biomarker, Responder) | Phase 2 Unfit: Glasdegib 100 mg+LDAC(Biomarker, Non-Responder)
Number analyzed (Participants) | 33 | 55
ratio | 1.60 [0.50 to 40.25] | 0.50 [0.03 to 20.60]

63. Secondary Outcome: Number of Participants With Corrected QT Interval Using Fridericia's Formula (QTcF) Values Meeting Predefined Criteria at Phase 1B
Description: Maximum absolute values and increases from baseline were summarized for QTcF interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula). Number of participants with QTcF meeting the following criteria is presented: QTcF interval:<450 msec; QTcF interval: 450 to <480 msec; QTcF interval: 480 to <500 msec; QTcF interval >=500 msec; QTcF interval increase from baseline: <30 msec; QTcF interval increase from baseline: 30 to <60 msec; QTcF interval increase from baseline >=60 msec. Arms in the time frame description are defined as: Arm A, Glasdegib +LDAC; Arm B, Glasdegib + Decitabine; Arm C, Glasdegib + Cytarabine/Daunorubicin. End of treatment in the time frame were defined as: maximum of 12 cycles from start of therapy or until disease progression or relapse, participant refusal or unacceptable toxicity occurred, whichever came first.
Time Frame: 1 year
Population: QTc analysis set: all participants enrolled in the study having at least 1 ECG assessment after receiving at least 1 dose of glasdegib.
Measure: Number; unit: Participants
Arm/Group | Phase 1B: Glasdegib + LDAC | Phase 1B: Glasdegib + Decitabine | Phase 1B: Glasdegib + Cytarabine/Daunorubicin
Number analyzed (Participants) | 21 | 7 | 22
Participants
  QTcF interval increase < 30 msec | 16 | 2 | 14
  QTcF interval increase: 30 to < 60 msec | 5 | 3 | 6
  QTcF interval increase >= 60 msec | 0 | 2 | 2
  Maximum QTcF interval < 450 msec | 10 | 4 | 10
  Maximum QTcF interval: 450 to < 480 msec | 11 | 2 | 10
  Maximum QTcF interval: 480 to < 500 msec | 0 | 0 | 1
  Maximum QTcF interval >= 500 msec | 0 | 1 | 1

64. Secondary Outcome: Number of Participants With Corrected QT Interval Using Fridericia's Formula (QTcF) Values Meeting Predefined Criteria at Phase 2 Fit and Unfit
Description: Maximum absolute values and increases from baseline were summarized for QTcF interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula). Number of participants with QTcF meeting the following criteria is presented:QTcF interval:<450 msec; QTcF interval: 450 to <480 msec; QTcF interval: 480 to <500 msec; QTcF interval >=500 msec; QTcF interval increase from baseline: <30 msec; QTcF interval increase from baseline: 30 to <60 msec; QTcF interval increase from baseline >=60 msec. End of treatment in the time frame were defined as: maximum of 12 cycles from start of therapy or until disease progression or relapse, participant refusal or unacceptable toxicity occurred, whichever came first.
Time Frame: 1 year
Population: as for outcome 63
Measure: Number; unit: Participants
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 68 | 83 | 17
Participants
  QTcF interval increase < 30 msec | 41 | 60 | 12
  QTcF interval increase: 30 to < 60 msec | 21 | 19 | 4
  QTcF interval increase >= 60 msec | 6 | 4 | 1
  Maximum QTcF interval < 450 msec | 46 | 46 | 8
  Maximum QTcF interval: 450 to < 480 msec | 18 | 29 | 4
  Maximum QTcF interval: 480 to < 500 msec | 3 | 3 | 3
  Maximum QTcF interval >= 500 msec | 1 | 5 | 2

65. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) at Phase 1B (All Causality)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event did not necessarily had a causal relationship with the treatment or usage. Treatment Emergent AEs were those with initial onset or increasing in severity after the first dose of study medication and occurred within 28 days post last dose. AEs were graded by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 : Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: 4 years
Population: Safety analysis set: all enrolled participants who received at least 1 dose of any of the study medications for each drug combination.
Measure: Number; unit: Participants
Arm/Group | Phase 1B: Glasdegib + LDAC | Phase 1B: Glasdegib + Decitabine | Phase 1B: Glasdegib + Cytarabine/Daunorubicin
Number analyzed (Participants) | 23 | 7 | 22
Participants
  Grade 1 AEs | 1 | 1 | 0
  Grade 2 AEs | 2 | 0 | 3
  Grade 3 AEs | 3 | 1 | 8
  Grade 4 AEs | 10 | 4 | 10
  Grade 5 AEs | 7 | 1 | 1
  Missing or unknown AEs | 0 | 0 | 0

66. Secondary Outcome: Number of Participants With Treatment-emergent AEs at Phase 1B (Treatment-related)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event did not necessarily had a causal relationship with the treatment or usage. Treatment Emergent AEs were those with initial onset or increasing in severity after the first dose of study medication and occurred within 28 days post last dose. Treatment-related AEs were AEs related to glasdegib and/or backbone chemotherapy. AEs were graded by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 : Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: 4 years
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | Phase 1B: Glasdegib + LDAC | Phase 1B: Glasdegib + Decitabine | Phase 1B: Glasdegib + Cytarabine/Daunorubicin
Number analyzed (Participants) | 23 | 7 | 22
Participants
  Grade 1 AEs | 3 | 2 | 2
  Grade 2 AEs | 2 | 0 | 7
  Grade 3 AEs | 7 | 0 | 3
  Grade 4 AEs | 6 | 4 | 10
  Grade 5 AEs | 3 | 0 | 0
  Missing or unknown AEs | 0 | 0 | 0

67. Secondary Outcome: Number of Participants With Treatment-emergent AEs Categorized by Seriousness at Phase 1B
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event did not necessarily had a causal relationship with the treatment or usage. Treatment Emergent AEs were those with initial onset or increasing in severity after the first dose of study medication and occurred within 28 days post last dose. An serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect.
Time Frame: 4 years
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin
Number analyzed (Participants) | 17 | 6 | 4 | 3 | 16 | 6
Participants
  AEs | 17 | 6 | 4 | 3 | 16 | 6
  SAEs | 13 | 5 | 4 | 2 | 10 | 3

68. Secondary Outcome: Number of Participants With Treatment-emergent AEs at Phase 2 Fit and Unfit (All Causality)
Description: as for outcome 65
Time Frame: 4 years
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 69 | 84 | 41
Participants
  Grade 1 AEs | 0 | 2 | 0
  Grade 2 AEs | 1 | 4 | 1
  Grade 3 AEs | 11 | 15 | 8
  Grade 4 AEs | 52 | 39 | 15
  Grade 5 AEs | 5 | 24 | 17
  Missing or unknown AEs | 0 | 0 | 0

69. Secondary Outcome: Number of Participants With Treatment-emergent AEs at Phase 2 Fit and Unfit (Treatment-related)
Description: as for outcome 66
Time Frame: 4 years
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 69 | 84 | 41
Participants
  Grade 1 AEs | 0 | 4 | 4
  Grade 2 AEs | 4 | 9 | 6
  Grade 3 AEs | 15 | 20 | 3
  Grade 4 AEs | 46 | 34 | 10
  Grade 5 AEs | 1 | 1 | 1
  Missing or unknown AEs | 0 | 0 | 0

70. Secondary Outcome: Number of Participants With Treatment-emergent AEs Categorized by Seriousness at Phase 2 Fit and Unfit
Description: as for outcome 67
Time Frame: 4 years
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
Number analyzed (Participants) | 69 | 84 | 41
Participants
  AEs | 69 | 84 | 41
  SAEs | 35 | 68 | 32

ADVERSE EVENTS:
Time Frame: 4 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. All-cause mortality reflects the number of deaths from start of treatment to and including 28 days after last dose. Safety analysis set was evaluated.
Arm/Group | Phase 1B: Glasdegib 100 mg + LDAC | Phase 1B: Glasdegib 200 mg + LDAC | Phase 1B: Glasdegib 100 mg + Decitabine | Phase 1B: Glasdegib 200 mg + Decitabine | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin | Phase 2 Unfit: Glasdegib 100 mg + LDAC | Phase 2 Unfit: LDAC Alone
All-Cause Mortality (participants affected / at risk) | 6/17 | 1/6 | 1/4 | 0/3 | 0/16 | 1/6 | 5/69 | 26/84 | 17/41
Serious Adverse Events (participants affected / at risk) | 13/17 | 5/6 | 4/4 | 2/3 | 10/16 | 3/6 | 35/69 | 68/84 | 32/41
Other Adverse Events (participants affected / at risk) | 16/17 | 6/6 | 4/4 | 3/3 | 16/16 | 6/6 | 69/69 | 82/84 | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1B: Glasdegib 100 mg + LDAC (N=17) | Phase 1B: Glasdegib 200 mg + LDAC (N=6) | Phase 1B: Glasdegib 100 mg + Decitabine (N=4) | Phase 1B: Glasdegib 200 mg + Decitabine (N=3) | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin (N=16) | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin (N=6) | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin (N=69) | Phase 2 Unfit: Glasdegib 100 mg + LDAC (N=84) | Phase 2 Unfit: LDAC Alone (N=41)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 1 | 1 | 1 | 14 | 24 | 7
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Disease progression (General disorders) | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 10 | 5
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 4 | 19 | 7
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 5
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar puncture abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bipolar II disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mydriasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laboratory test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic encephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urogenital infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1B: Glasdegib 100 mg + LDAC (N=17) | Phase 1B: Glasdegib 200 mg + LDAC (N=6) | Phase 1B: Glasdegib 100 mg + Decitabine (N=4) | Phase 1B: Glasdegib 200 mg + Decitabine (N=3) | Phase 1B: Glasdegib 100 mg + Cytarabine/Daunorubicin (N=16) | Phase 1B: Glasdegib 200 mg + Cytarabine/Daunorubicin (N=6) | Phase 2 Fit: Glasdegib 100 mg + Cytarabine/Daunorubicin (N=69) | Phase 2 Unfit: Glasdegib 100 mg + LDAC (N=84) | Phase 2 Unfit: LDAC Alone (N=41)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 1 | 4 | 1 | 28 | 37 | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 8 | 2 | 38 | 8 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 9 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 0 | 2 | 2 | 4 | 1 | 15 | 13 | 8
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1 | 2 | 1 | 3 | 2 | 23 | 26 | 11
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 7 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 5 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scleral pigmentation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 10 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 1 | 1 | 6 | 0 | 20 | 15 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 7 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 7 | 3 | 2 | 1 | 10 | 3 | 32 | 21 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 2 | 2 | 0 | 10 | 6 | 49 | 24 | 9
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 10 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 4 | 1 | 12 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 6 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 4 | 2 | 5 | 7 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 2 | 4
Nausea (Gastrointestinal disorders) | 6 | 4 | 4 | 1 | 14 | 3 | 40 | 30 | 5
Oral disorder (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 5 | 0 | 17 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 5 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 5 | 4 | 25 | 18 | 4
Asthenia (General disorders) | 3 | 1 | 1 | 2 | 1 | 0 | 8 | 10 | 8
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 9 | 1
Chills (General disorders) | 1 | 1 | 0 | 1 | 5 | 0 | 21 | 5 | 1
Fatigue (General disorders) | 6 | 1 | 1 | 2 | 6 | 2 | 25 | 26 | 8
Gait disturbance (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 8 | 6 | 2
Nodule (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 6 | 0 | 0
Oedema peripheral (General disorders) | 5 | 1 | 0 | 1 | 7 | 2 | 22 | 22 | 7
Pain (General disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 6 | 4 | 3
Performance status decreased (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 0 | 1 | 0 | 10 | 1 | 34 | 23 | 9
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Genital infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 2 | 1 | 6 | 9 | 3
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 8 | 5 | 5
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0 | 0 | 6 | 5 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 9 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 4 | 1 | 21 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 17 | 6 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 13 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 19 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 2 | 1 | 1 | 0 | 1 | 14 | 9 | 3
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 7 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 3 | 5
Karnofsky scale worsened (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 6 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 12 | 11 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 18 | 14 | 4
Weight decreased (Investigations) | 1 | 1 | 1 | 0 | 1 | 1 | 9 | 17 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 4 | 0 | 20 | 13 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 2 | 2 | 26 | 29 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 6 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 7 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 3 | 2 | 18 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 5 | 2 | 22 | 5 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 0 | 6 | 2 | 37 | 13 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 4 | 2 | 20 | 8 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 5 | 1 | 23 | 10 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 3 | 0 | 15 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 11 | 10 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 4 | 1 | 12 | 9 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 2 | 10 | 2 | 11 | 19 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 6 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 7 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 3 | 1 | 5 | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 4 | 3 | 9 | 15 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 1 | 2 | 12 | 18 | 4
Dysgeusia (Nervous system disorders) | 4 | 4 | 1 | 1 | 7 | 1 | 19 | 21 | 1
Headache (Nervous system disorders) | 3 | 1 | 1 | 0 | 9 | 2 | 22 | 11 | 5
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 0 | 3 | 1 | 15 | 3 | 4
Apathy (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 7 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0 | 0 | 1 | 2 | 4 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 0 | 5 | 0 | 19 | 10 | 2
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 3 | 2 | 8 | 7 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 5 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 1 | 1 | 2 | 14 | 18 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 3 | 2 | 13 | 21 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 3 | 1 | 11 | 7 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 8 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 12 | 9 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 9 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 4 | 2 | 16 | 9 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 7 | 2
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 11 | 7 | 4
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 10 | 6 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 3 | 1 | 14 | 11 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 9 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 12 | 6 | 1
Hypotension (Vascular disorders) | 1 | 2 | 0 | 0 | 4 | 0 | 14 | 12 | 4
Ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.